CLINICAL TRIAL: NCT00119743
Title: Assess, in Young Children, the Efficacy in Preventing Acute Otitis Media (AOM) of GSK Biologicals Undecavalent Pneumococcal-protein D Conjugate Vaccine, When Administered as a Three Dose Primary Vaccination Course During the First Year of Life With a Booster Dose in the Second Year of Life.
Brief Title: A Efficacy Against Otitis Media in Children With 11 Valent Pneumococcal Vaccine
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 347414/010
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis A
Keywords: Prophylaxis pneumococcal vaccine
MeSH Terms: conditions — Hepatitis A

INTERVENTIONS:
Biological: undecavalent pneumococcal-protein D conjugate vaccine

SUMMARY:
The purpose of this study is to assess the efficacy in young children in preventing acute otitis media due to vaccine serotype pneumococcal or non typable Hemophilus influenza, following immunization with an 11-valent pneumococcal vaccine according to a 3 dose primary vaccination in the first year of life, with booster dose in the second year of life. Prophylactic immunization with pneumococcal conjugate vaccine is compared to placebo (hepatitis A vaccine).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 6 weeks and 5 months (42-152 days) of age at the time of first vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.

Ages: 6 Weeks to 27 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5000
Dates: Start 2000-10; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
To demonstrate the efficacy of the 11 Pn-PD vaccine in preventing AOM caused by vaccine-type pneumococcus in fully vaccinated children less than 2 years of age.

SECONDARY OUTCOMES:
To assess the efficacy of the 11 Pn-PD vaccine in preventing AOM caused by NTHI in fully vaccinated children less than 2 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (35):
- Czechia (16):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, České Budějovice
  - GSK Investigational Site, Děčín
  - GSK Investigational Site, Fryštát
  - GSK Investigational Site, Frýdek-Místek
  - GSK Investigational Site, Havlíčkův Brod
  - GSK Investigational Site, Hlinsko
  - GSK Investigational Site, Jičín
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Litoměřice
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Ústí nad Labem
  - GSK Investigational Site, Znojmo
- Slovakia (19):
  - GSK Investigational Site, Dolný Kubín
  - GSK Investigational Site, Dubnica nad Váhom
  - GSK Investigational Site, Košťany nad Turcom
  - GSK Investigational Site, Liptovský Hrádok
  - GSK Investigational Site, Liptovský Mikuláš
  - GSK Investigational Site, Martin
  - GSK Investigational Site, Námestovo
  - GSK Investigational Site, Nitra
  - GSK Investigational Site, Nová Dubnica
  - GSK Investigational Site, Nové Mesto nad Váhom
  - GSK Investigational Site, Nové Zámky
  - GSK Investigational Site, Považská Bystrica
  - GSK Investigational Site, Púchov
  - GSK Investigational Site, Ružomberok
  - GSK Investigational Site, Sučany
  - GSK Investigational Site, Štúrovo
  - GSK Investigational Site, Šurany
  - GSK Investigational Site, Trenčín
  - GSK Investigational Site, Zlaté Moravce

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Poolman J, Kriz P, Feron C, Di-Paolo E, Henckaerts I, Miseur A, Wauters D, Prymula R, Schuerman L. Pneumococcal serotype 3 otitis media, limited effect of polysaccharide conjugate immunisation and strain characteristics. Vaccine. 2009 May 21;27(24):3213-22. doi: 10.1016/j.vaccine.2009.03.017. Epub 2009 Mar 26. PMID 19446194
- [Background] Poolman J, Frasch C, Nurkka A, Kayhty H, Biemans R, Schuerman L. Impact of the conjugation method on the immunogenicity of Streptococcus pneumoniae serotype 19F polysaccharide in conjugate vaccines. Clin Vaccine Immunol. 2011 Feb;18(2):327-36. doi: 10.1128/CVI.00402-10. Epub 2010 Dec 1. PMID 21123523
- [Background] Prymula R, Peeters P, Chrobok V, Kriz P, Novakova E, Kaliskova E, Kohl I, Lommel P, Poolman J, Prieels JP, Schuerman L. Pneumococcal capsular polysaccharides conjugated to protein D for prevention of acute otitis media caused by both Streptococcus pneumoniae and non-typable Haemophilus influenzae: a randomised double-blind efficacy study. Lancet. 2006 Mar 4;367(9512):740-8. doi: 10.1016/S0140-6736(06)68304-9. PMID 16517274
- [Background] Prymula R, Chlibek R, Splino M, Kaliskova E, Kohl I, Lommel P, Schuerman L. Safety of the 11-valent pneumococcal vaccine conjugated to non-typeable Haemophilus influenzae-derived protein D in the first 2 years of life and immunogenicity of the co-administered hexavalent diphtheria, tetanus, acellular pertussis, hepatitis B, inactivated polio virus, Haemophilus influenzae type b and control hepatitis A vaccines. Vaccine. 2008 Aug 18;26(35):4563-70. doi: 10.1016/j.vaccine.2008.05.080. Epub 2008 Jun 17. PMID 18602724
- [Background] Schuerman L, Prymula R, Henckaerts I, Poolman J. ELISA IgG concentrations and opsonophagocytic activity following pneumococcal protein D conjugate vaccination and relationship to efficacy against acute otitis media. Vaccine. 2007 Mar 1;25(11):1962-8. doi: 10.1016/j.vaccine.2006.12.008. Epub 2006 Dec 26. PMID 17258357
- [Background] Schuerman L, Prymula R, Chrobok V, Dieussaert I, Poolman J. Kinetics of the immune response following pneumococcal PD conjugate vaccination. Vaccine. 2007 Mar 1;25(11):1953-61. doi: 10.1016/j.vaccine.2006.12.007. Epub 2006 Dec 26. PMID 17258358
- [Background] Schuerman L, Borys D, Hoet B, Forsgren A, Prymula R. Prevention of otitis media: now a reality? Vaccine. 2009 Sep 25;27(42):5748-54. doi: 10.1016/j.vaccine.2009.07.070. Epub 2009 Aug 8. PMID 19666154
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 347414/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 347414/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 347414/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 347414/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 347414/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 347414/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register